CLINICAL TRIAL: NCT03586557
Title: Effectiveness of Plasma Exchange in Treating With Severe Acute AQP4-Ab Positive Optic Neuritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Wei Shihui, Professor of Neuro-Ophthalmology, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PETON
Record Dates: First submitted 2018-06-13; First posted 2018-07-13 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Optic Neuritis
Keywords: Optic Neuritis; aquaporin4-IgG; Treatment
MeSH Terms: conditions — Optic Neuritis | interventions — Plasma Exchange; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: a open-labeled randomized comparison study
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessor was masked to avoid measured bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid & Plasma Exchange (Experimental): 1000mg intravenous methylprednisolone daily for 3~5 days and subsequent taper, combined with plasma exchange every other day for five times in all
  Interventions: Device: Corticosteroid & Plasma exchange
- Corticosteroid (Active Comparator): 1000mg intravenous methylprednisolone daily for 3~5 days, and subsequent corticosteroid decrement.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Device: Corticosteroid & Plasma exchange — High-dose intravenous methylprednisolone 1000mg 3~5 days and subsequent taper, combined simultaneous plasma exchange 5 times in all
  Other Names: CS+PE
  Arms: Corticosteroid & Plasma Exchange
Drug: Corticosteroid — High-dose intravenous methylprednisolone 1000mg 3~5 days and subsequent taper
  Other Names: CS
  Arms: Corticosteroid

SUMMARY:
Patients aged between 18 and 70 with acute aquaporin-4 immunoglobulin G antibodies (AQP4-IgG) positive optic neuritis, irrespective of prior using of corticosteroids in this episode of disease, are chosen by the physician. Patients will then be randomized to receive high dose of intravenous corticosteroids combined with plasma exchange (PE), or merely high dose of intravenous corticosteroids followed subsequent taper. The main outcome of visual acuity and OCT parameters will be compared at baseline, one, three and six months after treatments, and other assessments will also be recorded and compared. This will allow for determination on whether additional PE plays a role in better prognosis in acute AQP4-IgG positive optic neuritis.

DETAILED DESCRIPTION:
Definition:

This will be a parallel designed, open-labeled, randomized add-on comparison study between 1) intravenous high dose corticosteroids combined with plasma exchange (PE) and 2) merely intravenous high dose corticosteroids followed subsequent taper of the improvement of optic nerve function in acute aquaporin-4 immunoglobulin G antibodies (AQP4-IgG) positive optic neuritis. The investigators will compare assessments at baseline with those at one, three and six months post treatments.

Patients:

Subjects will be recruited from in-patients who were diagnosed as AQP4-IgG positive optic neuritis in Neuro-Ophthalmology Department in People's Liberation of Army General Hospital (PLAGH) in Beijing, China.

Eligible participants should have inaugural or recurrent unilateral or bilateral optic neuritis attack(s) within 30 days from the first symptom onset. Only affected eyes with VA less than 20/200 at baseline will be included in the study. All of the participants have to have positive serum AQP4-IgG. Enrollment will be allowed irrespective of whether a previous diagnosis of neuromyelitis optica spectrum disorders (NMOSD) was made.

Participants will be randomly assigned (1:1) to exclusively intravenous corticosteroid (CS group) or sequential intravenous corticosteroid and PE( CS and PE group) .

All participants will receive intravenous corticosteroid (1g of methylprednisolone per day for 3~5days, and subsequent taper). The treatment will be started as soon as the participant is admitted to the hospital. The participants in CS and PE group will receive add-on five consecutive PE every other day performed in the ward.

Primary and secondary endpoints:

The primary endpoint will be the value of visual acuity (VA ) at end of follow-up (6 months) in the affected eyes. VA was assessed separately for each eye using Snellen's test chart at baseline, one, three and six months, and was converted to LogMAR for calculation of the mean visual acuity. If the patient has a relapse during the follow-up, the last VA recorded before the relapse will be the final VA outcome of the patient.

Optical Coherence Tomography (OCT) parameters assessed at months 6 will be another primary endpoint. OCT will be performed with spectrum domain OCT (SD-OCT) (Carl Zeiss 5000). Peripapillary retinal nerve fiber layer (pRNFL), macular retinal thickness and macular Ganglion Cell Layer + inner plexiform layer (mGCIPL) will be measured by one skilled technician at the condition of dilated pupil to avoid bias of measurement. Parameters above will be recorded thereafter.

Secondary endpoints will study the numbers of relapses during the follow-up of 6 months, optic nerve conduction velocity measured by Flash Visual Evoked Potential (FVEP) at the end of follow-up (6 months). FVEP will be recorded by visual electro-physiology equipment (Roland RETI-Port/Scan 21). The same technician will perform all the assessments for all the patients to avoid bias of measurement. A final latency assessment was analysed at study end.

Titer of serum AQP4-IgG within 1 month after their attack and six months after treatment will be recorded. Orbital MRI will be assessed and compared if it is necessary.

Security indexes:

Safety assessment at screening，baseline，one , three, and six month are: physical examination and vital signs including blood pressure (BP), heart rate (HR). Hematology and blood chemistry will be assessed as well. blood routine test, coagulation Test, and serum electrolyte will be tested during the PE treatment and followed up at one, three and six months. Allergies during PE treatment will be recorded by doctors. Patients experiencing severe adverse events would be remove from the treatment arm. However, patients with slight or medium adverse events should complete their PE treatment unless they require to quit.

Sample size:

The estimated mean VA outcome of AQP4-IgG positive optic neuritis 6 months after its attack is expected to be about 1.4 (LogMAR) with its standard deviation (SD) around 1.3 (LogMAR), based on 2 observation reports. Another observational study found that mean VA outcome after PE combined corticosteroid treated AQP4-IgG positive optic neuritis was 0.75 (LogMAR). The investigators assume that to achieve 80% power at 5% significance level, using a parallel design, the sample size needs to be 64 cases per group and 128 in all. By accounting for 10% patients potentially withdrawing consent or being lost to follow-up over the course of the study, the final sample size will be increased to 71 cases per arm and 142 patients in all.

Planned Statistical Analysis:

The primary analysis will be intention-to-treat. The outcome of the superiority clinical trial will be assessed based on a two-sided 95% confidence interval around the mean VA and OCT outcome, showing a credible range for true difference between merely corticosteroid and corticosteroid combined PE treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 70 years old
2. Serum AQP4-IgG positive optic neuritis
3. Patients must have their VA less than 20/200
4. Course of disease is less than 1 month
5. Patients must provide written informed consent

Exclusion Criteria:

1. Females who are pregnancy
2. Patients who are severely allergic to plasma or albumin
3. Patients who have systemic disease and can not accept PE
4. Patients with a tendency to thrombus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity (LogMAR) | from baseline to 6 months
  the differences in Visual Acuity outcomes between treatment arm and control arm
Change in OCT parameters over time | baseline to 6 months
  Difference in mean thickness of peripapillary retinal nerve fiber layer and macular Ganglion Cell Complex between treatment group and control group

SECONDARY OUTCOMES:
Change in Flash Visual Evoked Potential over time | baseline to 6 month
  Difference in P2 peak time and value between treatment group and control group
rate of recurrence over time | baseline to 6 months
  the differences in rate of recurrence (number of recurrence patients / number of patients in their arms) between treatment group and control group
change in serum AQP4-IgG titer over time | baseline to 6 months
  compare the different changes in serum AQP4-IgG titer (before treatment and 6 months follow-up) between PE combined corticosteroid group and only corticosteroid group
orbital MRI | baseline to 6 months
  orbital MRI will be assessed if it is necessary

OTHER OUTCOMES:
Blood Pressure | baseline, during PE treatment and followed up at one, three and six months
  the change of Blood Pressure at baseline, during PE treatment and follow up
Heart Rate | baseline, during PE treatment and followed up at one, three and six months
  the change of Heart Rate at baseline, during PE treatment and follow up
Rooting Blood Test | baseline, during PE treatment and followed up at one, three and six months
  the change of Rooting Blood Test outcome at baseline, during PE treatment and follow up
Coagulation test | baseline, during PE treatment and followed up at one, three and six months
  the change of Coagulation test outcome at baseline, during PE treatment and follow up
Serum electrolyte | baseline, during PE treatment and followed up at one, three and six months
  the change of Serum electrolyte at baseline, during PE treatment and follow up
side effects | baseline to 6 months
  record the side effects during the period of PE treatment

CONTACTS AND LOCATIONS:
Overall Officials: Quangang Xu, PhD, Principal Investigator — Chinese PLA General Hospital; Huanfen Zhou, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- People's Liberation of Army General Hospital (PLAGH), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No